CLINICAL TRIAL: NCT02575105
Title: Bispectral Index Monitoring of Propofol Anesthesia in Patients With Hydrocephalus. A Prospective Observational Study
Brief Title: BIS Monitoring of Patients With Hydrocephalus
Acronym: BIS1
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Collaborators: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Ashraf Dahaba, MD, Doz. Dr., Suez Canal University
Other Study IDs: MUGraz
Record Dates: First submitted 2015-10-10; First posted 2015-10-14 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Hydrocephalus
Keywords: Bispectral Index Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pediatric Hydrocephalus: In the first study 15 pediatric patients with hydrocephaly and 15 pediatric control patients at approximately the same age group will be included in the study.
- Pediatric Control: In the first study 15 pediatric patients with hydrocephaly and 15 pediatric control patients at approximately the same age group will be included in the study.
- Adult Hydrocephalus: In the second study 15 post cerebral hemorrhage adult patients undergoing ventriculo-peritoneal shunt placements and 15 adult control patients will be included in the study
- Adult Control: In the second study 15 post cerebral hemorrhage adult patients undergoing ventriculo-peritoneal shunt placements and 15 adult control patients will be included in the study

SUMMARY:
We tested the hypothesis that BIS values are altered in pediatric patients with hydrocephaly. We also tested the hypothesis that BIS values are altered in adult post cerebral hemorrhage patients with hydrocephaly undergoing ventricular-peritoneal shunt placement

DETAILED DESCRIPTION:
Context: Enlarged skull circumference in patients with hydrocephalus might alter bispectral index (BIS) values; as distorted skull contour distances sensors from a shifted cerebral mass as well as mental dysfunction as a result of disrupted Cerebrospinal fluid circulation.

Objectives: Investigators tested the hypothesis that BIS values are altered in pediatric patients with hydrocephaly. Investigators also tested the hypothesis that BIS values are altered in adult post cerebral hemorrhage patients with hydrocephaly undergoing ventricular-peritoneal shunt placement.

Methods: After ethics committee approval participants, or their next of kin, who gave written informed consent were recruited in the study. Investigators excluded potential participants suffering from hepatic disease. In the first study 15 pediatric patients with hydrocephaly and 15 pediatric control patients at approximately the same age group were included in the study.

In the second study 15 post cerebral hemorrhage adult patients undergoing ventricular-peritoneal shunt placements and 15 adult control patients were included in the study.

2 BIS sensors were placed on patients' forehead and connected to BIS-Vista monitors. In a quiet anesthesia induction room investigators recorded BIS-Vista for 10 min before induction.

Remifentanil 4 ng ml-1 was started and propofol TCI was kept constant at 4 microg ml-1 with no adjustments for a 1 h anesthesia maintenance study-recording period when time of surgery allowed. Investigators also noted BIS values immediately before and after a patent ventricular-peritoneal shunt was successfully installed. After conclusion of surgical procedures, remifentanil and propofol infusions were terminated and this marked the beginning of the recovery phase of the study where we recorded BIS values for another 20 min emergence from anesthesia.

ELIGIBILITY:
Inclusion Criteria: . In the first study 15 pediatric patients with hydrocephaly and 15 pediatric control patients at approximately the same age group will be included in the study.

In the second study 15 post cerebral hemorrhage adult patients undergoing ventriculo-peritoneal shunt placements and 15 adult control patients will be included in the study.

Exclusion Criteria: Patients with Liver disease

Ages: 1 Month to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: . In the first study 15 pediatric patients with hydrocephaly and 15 pediatric control patients at approximately the same age group will be included in the study.
  In the second study 15 post cerebral hemorrhage adult patients undergoing ventriculo-peritoneal shunt placements and 15 adult control patients will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Difference in Bispectral Index Value | Duration of Surgical Operation
  Might be statistically different

REFERENCES:
- [Background] Dahaba AA. Different conditions that could result in the bispectral index indicating an incorrect hypnotic state. Anesth Analg. 2005 Sep;101(3):765-773. doi: 10.1213/01.ane.0000167269.62966.af. PMID 16115989
- [Background] Dahaba AA, Worm HC, Zhu SM, Bao FP, Salah A, Zakaria S, Bornemann H, Stadlbauer V, Rehak PH, Metzler H, Stauber RE. Sensitivity and specificity of bispectral index for classification of overt hepatic encephalopathy: a multicentre, observer blinded, validation study. Gut. 2008 Jan;57(1):77-83. doi: 10.1136/gut.2007.129130. Epub 2007 Aug 14. PMID 17698861
- [Background] Dahaba AA, Xue JX, Zhao GG, Liu QH, Xu GX, Bornemann H, Rehak PH, Metzler H. BIS-vista occipital montage in patients undergoing neurosurgical procedures during propofol-remifentanil anesthesia. Anesthesiology. 2010 Mar;112(3):645-51. doi: 10.1097/ALN.0b013e3181cf4111. PMID 20179501
- [Background] Dahaba AA, Lin H, Ye XF, Lin J, Zhang N, Lian QQ. Bispectral index monitoring of propofol anesthesia in pediatric patients with hydrocephalus. A prospective observational study. Paediatr Anaesth. 2014 Nov;24(11):1190-2. doi: 10.1111/pan.12508. No abstract available. PMID 25279677